CLINICAL TRIAL: NCT03751306
Title: Sensory-Motor and Cardiorespiratory Rehabilitation Associated With Transcranial Laser Therapy in Patients With Central Nervous System Injury
Brief Title: Aerobic Exercise and Transcranial Low Laser Therapy in Patients With Central Nervous System Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade do Vale do Paraíba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 94858718.3.0000.5503
Record Dates: First submitted 2018-11-01; First posted 2018-11-23 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Post Stroke; Post-Traumatic Headache; Spinal Injuries; Cerebral Palsy, Spastic; Surgery; Sclerosis, Multiple; Spastic
Keywords: Neurological Diseases; Cardiorespiratory Rehabilitation; Aerobic exercise; Fotobiomodulação Transcraniana
MeSH Terms: conditions — Post-Traumatic Headache; Spinal Injuries; Cerebral Palsy; Multiple Sclerosis; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control-Cardiorespiratory Rehabilitation (Active Comparator): These individuals will compose the control group for transcranial laser therapy, which will only receive cardiorespiratory rehabilitation.
  Interventions: Procedure: Cardiorespiratory Rehabilitation
- Transcranial Photobiomodulation Placebo (Placebo Comparator): In this group, the application of laser irradiation will be simulated, and the laser will be turned off. And the simulation of irradiation, the individuals will initiate cardiorespiratory rehabilitation.
  Interventions: Procedure: Transcranial Photobiomodulation (Placebo); Procedure: Cardiorespiratory Rehabilitation
- Transcranial Photobiomodulation (Experimental): In this group, low-intensity irradiation will be applied and after irradiation, the volunteers will begin cardiorespiratory rehabilitation.
  Interventions: Procedure: Transcranial Photobiomodulation; Procedure: Cardiorespiratory Rehabilitation

INTERVENTIONS:
Procedure: Transcranial Photobiomodulation — Photobiomodulation Rehabilitation:
  Diode laser, λ infrared = 810 nm, 0.028 cm2 beam area, 100 mW power, 3.5 W / cm2 power density, 3 Joules / dot and Energy Density of 107.1 J / cm2). Each point will be radiated for 30 seconds. The regions of irradiation will be in the middle cerebral arteries (points F7 and F8 will be used as reference point according to the International System 10-20 of the electroencephalogram) and anterior cerebral artery (AFz point according to the International System 10-20 of the electroencephalogram) .
  Arms: Transcranial Photobiomodulation
Procedure: Transcranial Photobiomodulation (Placebo) — Photobiomodulation Placebo Therapy:
  The same apparatus of the transcranial group photobiomodulation and the same irradiation points will be used. However, during the procedure, with the laser off.
  Arms: Transcranial Photobiomodulation Placebo
Procedure: Cardiorespiratory Rehabilitation — Cardiorespiratory Rehabilitation:
  Aerobic training on the treadmill will be reliated for 30 minutes using the support of the Rehabilitation and Physical Activity Station BrainMov® (equipment with 4 pillars condition that favors the suspension and stabilization of people with neuromuscular dysfunctions of mild to severe impairment. For monitoring, the training heart rate equation - Karvonen equation, effort perception scale - BORG, systemic arterial pressure, peripheral oxygen saturation, and patient signs and symptoms will be used. Subsequently, respiratory exercises and muscle strengthening of lower limbs, final relaxation and general guidelines will be performed for research volunteer and his / her relatives.

SUMMARY:
Objective of this protocol will be to evaluate the parameters related to the function of the musculoskeletal and cardiorespiratory system, through a rehabilitation and training program for people with acquired central nervous system and multiple sclerosis. The study will consist of volunteers with acquired CNS lesions and multiple sclerosis of both sexes, between 18 and 85 years old, and who wander with or without aid devices, randomly divided into 3 groups: Group 1 (cardiopulmonary treatment), Group 2 (cardiopulmonary treatment and transcranial photobiomodulation application) and Group 3 (cardiopulmonary treatment and placebo laser). All groups will receive aerobic training on a treadmill (Moviment®) with the aid of a suspension equipment (BrainMov® Physical Activity Station). The transcranial photobiomodulation (laser diode, λ = 810 nm, beam area 0.028 cm², power of 100 mW, power density of 3.5 mW / cm², energy of 3 Joules / point and energy density of 107.1 J / cm2) will be applied on the skin / scalp and the International System 10-20 at points F7, F8 and AFz will be used as reference for irradiation. Muscular activation, heart rate variability, lung volumes and capacities, fatigability, exercise tolerance, cognition and quality of life will be evaluated before, during, at the end and after two months of rehabilitation. The treatment proposed in this study, using transcranial photobiomodulation, is expected to improve muscle, sensory, cardiorespiratory, cognitive functions and to interfere positively in the quality of life of the volunteers.

DETAILED DESCRIPTION:
Central nervous system (CNS) diseases can be acquired (such as stroke, spinal cord injury, and traumatic brain injury) or non-acquired (such as multiple sclerosis). Many diseases that affect the CNS can be fatal or cause sequelae, which affect the sensorimotor, cardiorespiratory and the quality of life of the individual. Subjects with neurological lesions present low resistance to exercise, a factor that can be attributed to decreased muscle recruitment, oxidative and metabolic capacity reduction, low aerobic resistance and increased energy expenditure. With that in mind, treatment proposals such as aerobic training and gait training with or without weight loss can maximize and restore the individual's functional abilities through active learning. Cardiorespiratory fitness in this patient profile has benefits in terms of fatigue retardation, gait improvement and regulation of the autonomic nervous system. Aerobic exercises change the heart rhythm, increase vascularity and provide oxygen. The association of these factors promote cerebral neuroprotective effect, stimulate the production of endogenous neutrotransmitters related to general well-being and favor neuroplasticity. Low-intensity laser therapy, especially transcranial photobiomodulation, has shown benefits in animals and humans such as cognitive and memory improvement, improvement in the behavioral picture, such as attenuation of depression and anxiety, and cortical oxygenation.

The study design is a randomized, double-blind, placebo-controlled trial that will compare the effect of cardiorespiratory rehabilitation, cardiorespiratory rehabilitation and low-intensity laser therapy, cardiorespiratory rehabilitation and placebo laser. It is worth mentioning that the use of a Placebo Therapy is restricted to Low Power Laser irradiation. This means that the three experimental groups will effectively be treated with cardiorespiratory rehabilitation, a therapy that improves physical fitness. The treatment with transcranial photobiomodulation irradiation aims to verify the effects and aggregates greater beneficial to the volunteers. In this case, the magnitude of the laser effect must be calculated by the difference (if any) of the group treated with "cardiorespiratory rehabilitation + laser" subtracted from the group treated with "cardiorespiratory rehabilitation + laser Placebo".

ELIGIBILITY:
Inclusion Criteria:

* Persons with stroke, traumatic brain injury, spinal cord trauma, post-operative brain tumor, chronic non-progressive encephalopathy and multiple sclerosis;
* Chronic neurological diseases, from 6 months of injury;
* Caucasian individuals;
* Age between 18 and 85 years;
* Both sexes;
* Individuals with the cognitive preserved;
* Persons who are able to wander on the treadmill voluntarily or through assistance from the Rehabilitation and Physical Activity Station BrainMov®;
* Persons who make continuous and regular use of medications prescribed by the physician for the control and / or treatment of chronic diseases;
* People with the release of the cardiologist for rehabilitation.

Exclusion Criteria:

* People who do not meet the inclusion criteria;
* Active smokers;
* Carriers of chronic respiratory diseases, such as COPD, asthma and bronchiectasis;
* Patients with decompensated heart disease;
* Obesity grade II - body mass index greater than 34.99 kg / m2;
* Patients with spinal cord injury above T6, who present autonomic dysreflexia;
* Patients with ASA A or B spinal cord injury;
* Patients with multiple sclerosis who are in an outbreak period;
* Patients taking betablockers;
* Hemorrhagic stroke.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-01-14 (Estimated); Primary Completion 2019-07-31 (Estimated); Study Completion 2020-03-05 (Estimated)

PRIMARY OUTCOMES:
Change in Muscular electrical activity (Surface electromyograph). | Baseline (before starting rehabilitation) and after 9 weeks.
  The surface electrodes will be positioned in the rectus femoris and femoral biceps muscles. The evaluation of the muscles will be realized during the squat movement. 10 seconds of signal collection (in triplicate).
Change in analysis of bipodal balance during the squat movement. | Baseline (before starting rehabilitation) and after 9 weeks.
  The balance evaluation will be performed during the squat movement on the power platform (Stabilometric analysis in Kgf). 10 seconds of signal collection (in triplicate).
Change in analysis of the heart rate variability to study the responses of the autonomic nervous system | Baseline (First day of rehabilitation) and after 9 weeks (Last day of rehabilitation).
  Heart rate variability will be assessed during aerobic training on the treadmill for 40 minutes (5 minutes of initial rest, 30 minutes of exercise and 5 minutes of final rest).
Change in Pulmonary function analysis (spirometry): forced vital capacity | Baseline (before starting rehabilitation) and after 9 weeks.
  Using the spirometry technique, forced vital capacity (measured in liters) will be evaluated. The volunteer will be asked to perform the maximum inspiration and exhale with maximum effort.
Change in Pulmonary function analysis (spirometry): forced expiratory volume in the first second | Baseline (before starting rehabilitation) and after 9 weeks.
  Using the spirometry technique, forced expiratory volume in the first second (measured in liters) will be evaluated. The volume of exhaled air in the first second in the forced vital capacity maneuver will be evaluated.
Change in Pulmonary function analysis (spirometry): Tiffeneau Index | Baseline (before starting rehabilitation) and after 9 weeks.
  Using the spirometry technique, Tiffeneau Index will be evaluated. The Tiffeneau index is the result of the division of forced expiratory volume in the first second in relation to forced vital capacity.
Change in Pulmonary function analysis (spirometry): maximum voluntary ventilation | Baseline (before starting rehabilitation) and after 9 weeks.
  Using the spirometry technique, maximum voluntary ventilation will be evaluated. Maximum voluntary ventilation is the largest volume of air that the individual can mobilize in one minute with maximum voluntary effort. The test gives an overview of the ventilatory function (measured in L / min).
Change in analysis of inspiratory muscle strength | Baseline (before starting rehabilitation) and after 9 weeks.
  The inspiratory muscle strength will be evaluated by means of the manovacuometer.
Analysis of expiratory muscle strength | Baseline (before starting rehabilitation) and after 9 weeks.
  The expiratory muscle strength will be evaluated by means of the manovacuometer
Change in analysis of Peak expiratory flow. | Baseline (before starting rehabilitation) and after 9 weeks.
  To analyze the velocity of the air out of the lungs.
Change in analysis of the thoracic expandability (axillary level). | Baseline (before starting rehabilitation) and after 9 weeks.
  In order to analyze the chest expansion at the axillary level, a metric tape placed at the torarico-axillary level will be used, which will measure the inspiratory and expiration mobility values, and will be subtracted (Insp-Exp).
Change in analysis of the thoracic expandability (xiphoid level). | Baseline (before starting rehabilitation) and after 9 weeks.
  In order to analyze the chest expansion at the xiphoid level, a metric tape will be used, placed at the thoracic-xiphoid level, which will measure the inspiratory and expiration mobility values and then be subtracted (Insp-Exp).
Change in analysis of abdominal level expandability. | Baseline (before starting rehabilitation) and after 9 weeks.
  In order to analyze abdominal expansibility, a tape measure will be used, placed at the level of the umbilical scar, which will measure the inspiratory and expiration mobility values and will be subtracted (Insp-Exp).
Change in analysis of change in Infrared Thermography. | Baseline (before starting rehabilitation) and after 9 weeks.
  By means of an infrared thermographic camera, the blood circulation of the lower limbs will be evaluated by the temperature difference.
Change in aariation of blood lactate level. | Baseline (before starting rehabilitation) and after 9 weeks.
  The blood lactate level will be measured by a lactometer, which will be collected from the volunteer's blood sample before starting the aerobic training on the treadmill and after training.
Change in 6-Minute Walk Test (Adapted) | Baseline (before starting rehabilitation) and after 9 weeks.
  The 6-minute-walk test will be adapted for neurological patients, which will be evaluated for exercise tolerance using a treadmill (Moviment RT200®). Volunteers will be assisted by the BrainMov® Rehabilitation and Physical Activity Station to stabilize the trunk and thus remain upright to wander on the treadmill
Change in Mini-Mental State Examination (MINI MENTAL). | Baseline (before starting rehabilitation) and after 9 weeks.
  To evaluate the cognitive functions, the MINI MENTAL test will be applied.
Change in Short Form 36 questionnaire (SF-36) | Baseline (before starting rehabilitation) and after 9 week.
  To evaluate the domains of quality of life: Functional Capacity, physical aspect, pain, general health, vitality, social aspect, emotional spectrum and mental health

SECONDARY OUTCOMES:
Follow-up: Evaluation Muscular electrical activity (Surface electromyograph) | The follow-up revaluation will be 2 months after the end of rehabilitation.
  Evaluation of muscular electrical activity after 9 weeks of the end of rehabilitation. The surface electrodes will be positioned in the rectus femoris and femoral biceps muscles. The evaluation of the muscles will be realized during the squat movement. 10 seconds of signal collection (in triplicate).
Follow-up: Analysis of bipodal balance during the squat movement | The follow-up revaluation will be 2 months after the end of rehabilitation.
  The balance evaluation will be performed during the squat movement on the power platform. 10 seconds of signal collection (in triplicate).
Follow-up: Analysis of the heart rate variability to study the responses of the autonomic nervous system | The follow-up revaluation will be 2 months after the end of rehabilitation.
  The heart rate variability will be evaluated during aerobic training on the treadmill using a frequency for 5 minutes of initial rest, 30 minutes of exercise and 5 minutes of final rest.
Follow-up: Pulmonary function analysis (spirometry): forced vital capacity | The follow-up revaluation will be 2 months after the end of rehabilitation.
  Using the spirometry technique, forced vital capacity (measured in liters) will be evaluated. The patient will be asked to perform the maximum inspiration and exhale with maximum effort.
Follow-up: Pulmonary function analysis (spirometry): forced expiratory volume in the first second | The follow-up revaluation will be 2 months after the end of rehabilitation.
  Using the spirometry technique, forced expiratory volume in the first second (measured in liters) will be evaluated. The volume of exhaled air in the first second in the forced vital capacity maneuver will be evaluated.
Follow-up: Pulmonary function analysis (spirometry):Tiffeneau Index | The follow-up revaluation will be 2 months after the end of rehabilitation.
  Using the spirometry technique, Tiffeneau Index will be evaluated. The Tiffeneau index is the result of the division of forced expiratory volume in the first second in relation to forced vital capacity.
Follow-up: Pulmonary function analysis (spirometry): maximum voluntary ventilation | The follow-up revaluation will be 2 months after the end of rehabilitation.
  Using the spirometry technique, maximum voluntary ventilation will be evaluated. Maximum voluntary ventilation is the largest volume of air that the individual can mobilize in one minute with maximum voluntary effort. The test gives an overview of the ventilatory function (measured in L / min).
Follow-up: Analysis of inspiratory muscle strength | The follow-up revaluation will be 2 months after the end of rehabilitation.
  The inspiratory muscle strength will be evaluated by means of the manovacuometer.
Follow-up: Analysis of expiratory muscle strength | The follow-up revaluation will be 2 months after the end of rehabilitation.
  The expiratory muscle strength will be evaluated by means of the manovacuometer.
Follow-up: Analysis of Peak expiratory flow. | The follow-up revaluation will be 2 months after the end of rehabilitation.
  To analyze the velocity of the air out of the lungs.
Follow-up: Analysis of the thoracic expandability (axillary level). | The follow-up revaluation will be 2 months after the end of rehabilitation.
  In order to analyze the chest expansion at the axillary level, a metric tape placed at the torarico-axillary level will be used, which will measure the inspiratory and expiration mobility values, and will be subtracted (Insp-Exp).
Follow-up: Analysis of the thoracic expandability (xiphoid level). | The follow-up revaluation will be 2 months after the end of rehabilitation.
  In order to analyze the chest expansion at the xiphoid level, a metric tape will be used, placed at the thoracic-xiphoid level, which will measure the inspiratory and expiration mobility values and then be subtracted (Insp-Exp).
Follow-up: Analysis of abdominal level expandability. | The follow-up revaluation will be 2 months after the end of rehabilitation.
  In order to analyze abdominal expansibility, a tape measure will be used, placed at the level of the umbilical scar, which will measure the inspiratory and expiration mobility values and will be subtracted (Insp-Exp).
Follow-up: Analysis of change in Infrared Thermography. | The follow-up revaluation will be 2 months after the end of rehabilitation.
  By means of an infrared thermographic camera, the blood circulation of the lower limbs will be evaluated by the temperature difference.
Follow-up: Variation of blood lactate level. | The follow-up revaluation will be 2 months after the end of rehabilitation.
  The blood lactate level will be measured by a lactometer, which will be collected from the volunteer's blood sample before starting the aerobic training on the treadmill and after training.
Follow-up: Analysis 6-Minute Walk Test (Adapted) | The follow-up revaluation will be 2 months after the end of rehabilitation.
  The 6-minute-walk test will be adapted for neurological patients, which will be evaluated for exercise tolerance using a treadmill (Moviment RT200®). Volunteers will be assisted by the BrainMov® Rehabilitation and Physical Activity Station to stabilize the trunk and thus remain upright to wander on the treadmill.
Follow-up: Evaluation Mini-Mental State Examination (MINI MENTAL). | The follow-up revaluation will be 2 months after the end of rehabilitation.
  To evaluate the cognitive functions, the MINI MENTAL test will be applied.
Follow-up: Evaluation Short Form 36 questionnaire (SF-36) | The follow-up revaluation will be 2 months after the end of rehabilitation.
  To evaluate the domains of quality of life: Functional Capacity, physical aspect, pain, general health, vitality, social aspect, emotional spectrum and mental health

CONTACTS AND LOCATIONS:
Overall Officials: Mário Oliveira Lima, Doctor, Principal Investigator — Universidade do Vale do Paraíba - Univap
Locations (1):
- Universidade do Vale do Paraíba, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pinto AP, Guimaraes CL, Souza GADS, Leonardo PS, Neves MFD, Lima FPS, Lima MO, Lopes-Martins RAB. Sensory-motor and cardiorespiratory sensory rehabilitation associated with transcranial photobiomodulation in patients with central nervous system injury: Trial protocol for a single-center, randomized, double-blind, and controlled clinical trial. Medicine (Baltimore). 2019 Jun;98(25):e15851. doi: 10.1097/MD.0000000000015851. PMID 31232920